CLINICAL TRIAL: NCT00052208
Title: A Phase I/II Study of an Oral Epidermal Growth Factor Receptor Tyrosine Kinase Inhibitor (EGFR-TKI), ZD 1839 (Iressa), [NSC #715055] With Radiation Therapy in Glioblastoma Multiforme
Brief Title: Gefitinib and Radiation Therapy in Treating Patients With Glioblastoma Multiforme
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2013-00849; RTOG-0211; CDR0000069330; RTOG-BR-0211; U10CA021661 (NIH)
Record Dates: First submitted 2003-01-24; First posted 2003-01-27 (Estimated); Last update posted 2020-10-30 (Actual); Status verified 2020-10

CONDITIONS: Adult Giant Cell Glioblastoma; Adult Glioblastoma; Adult Gliosarcoma
MeSH Terms: conditions — Glioblastoma; Gliosarcoma | interventions — Gefitinib; Radiotherapy; Radiation

ARMS (1):
- Treatment (gefitinib, radiation therapy) (Experimental): Patients receive gefitinib PO QD for 7 weeks. Beginning 1 week after initiation of gefitinib, patients undergo radiation therapy QD 5 days a week for 6 weeks. Treatment with gefitinib continues for up to 18 months in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: gefitinib; Radiation: radiation therapy; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: gefitinib — Given PO
  Other Names: Iressa; ZD 1839
Radiation: radiation therapy — Undergo radiation therapy
  Other Names: irradiation; radiotherapy; therapy, radiation
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase I/II trial studies the side effects and best dose of gefitinib when given together with radiation therapy and to see how well it works in treating patients with glioblastoma multiforme. Gefitinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Radiation therapy uses high energy x rays to kill tumor cells. Giving gefitinib together with radiation therapy may be an effective treatment for glioblastoma multiforme.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To identify the maximum tolerated dose of ZD 1839 (gefitinib) when given concurrently with cranial radiotherapy.

II. To determine if ZD 1839, given orally on a daily basis starting at the time of conventional radiation therapy (RT), may improve the overall survival of adults with newly-diagnosed supratentorial glioblastoma multiforme, compared with historical controls, stratifying by epidermal growth factor receptor (EGFR) status.

III. To determine, in a multi-institutional setting, the feasibility and toxicity of prescribing ZD 1839.

SECONDARY OBJECTIVES:

I. Whether ZD 1839 also improves progression-free survival in these patients.

OUTLINE: This is a phase I, dose-escalation study of gefitinib followed by a phase II study.

Patients receive gefitinib orally (PO) once daily (QD) for 7 weeks. Beginning 1 week after initiation of gefitinib, patients undergo radiation therapy QD 5 days a week for 6 weeks. Treatment with gefitinib continues for up to 18 months in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 4 months for 1 year, every 6 months for 2 years, and annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Histopathologically confirmed glioblastoma multiforme (with areas of necrosis)
* Diagnosis must be made by surgical biopsy or excision
* The tumor must be supratentorial in location
* The patient must have recovered from the effects of surgery, post-operative infection, or other complications before study entry
* Radiotherapy must begin =< five weeks after surgery, and Iressa (gefitinib) must begin one week prior to radiotherapy
* Patients must have an estimated survival of at least 8 weeks
* Zubrod performance status of 0-1
* A diagnostic contrast-enhanced magnetic resonance imaging (MRI) or computed tomography (CT) scan must be performed preoperatively and postoperatively prior to the initiation of radiotherapy; preoperative and postoperative scans must be the same type
* Patients diagnosed only by stereotactic biopsy do not require the postoperative scan
* Patients unable to undergo magnetic resonance (MR) imaging because of non-compatible devices can be enrolled, provided pre and postoperative CT scans are obtained and are of sufficient quality
* Hemoglobin >= 10 grams
* Absolute neutrophil count >= 1500 (ANC) per mm^3
* Platelets >= 100,000 per mm^3
* Blood urea nitrogen (BUN) =< 25 mg
* Creatinine =< 1.5 mg
* Bilirubin =< 2.0 mg
* Serum glutamate pyruvate transaminase (SGPT) or serum glutamic oxaloacetic transaminase (SGOT) =< 2 x normal range
* Patients must consent to submission of their tissue/serum
* The patient must sign a study-specific informed consent prior to study entry; if the patient's mental status precludes his/her giving informed consent, written informed consent may be given by the responsible family member

Exclusion Criteria:

* Recurrent or multifocal malignant gliomas
* Metastases detected below the tentorium or beyond the cranial vault
* Major medical illnesses or psychiatric impairments which, in the investigator's opinion, will prevent administration or completion of protocol therapy
* Previous radiotherapy to the head or neck (except for T1 glottic cancer), resulting in overlap of radiation fields
* Active connective tissue disorders, such as lupus or scleroderma which, in the opinion of the treating physician, may put the patient at high risk for radiation toxicity
* Previous malignancies, except for non-melanomatous skin cancers and carcinoma in situ of the uterine cervix or bladder, unless disease-free for >= 3 years
* Prior chemotherapy or radiosensitizers for cancers of the head and neck region
* Patients with known acquired immune deficiency (AIDS); patients with AIDS require complex therapeutic regimens; the pharmacokinetic interactions of these regimens with ZD 1839 are unknown and therefore, pose a safety risk related to excess toxicity or interference with anti-viral effectiveness
* Patients with known multiple sclerosis, as these patients may have decreased tolerance for radiation therapy to the brain
* Pregnant or lactating women, due to possible adverse effects on the developing fetus or infant due to study drug
* Patients treated on any other clinical protocols within 30 days prior to study entry or during participation in the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2002-03; Primary Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of gefitinib defined as the dose at which no patients develop acute grade 5 toxicity and less than 30% of patients developed acute dose limiting toxicity graded by the National Cancer Institute Common Toxicity Criteria v2.0 | Within 90 days from the start of radiotherapy treatment
Rate of late toxicities associated with gefitinib and standard cranial radiation, graded according to the NCI CTC v2.0 | Up to 10 years
Overall survival, by EGFR status | Up to 10 years

SECONDARY OUTCOMES:
Progression-free survival | Up to 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Arnab Chakravarti, Principal Investigator — Radiation Therapy Oncology Group
Locations (1):
- Radiation Therapy Oncology Group, Philadelphia, Pennsylvania, United States